CLINICAL TRIAL: NCT02137512
Title: Pilot Study 3 of Outpatient Control-to-Range: Safety and Efficacy With Day-and-Night In-Home Use
Acronym: CTR3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pilot 3 Outpatient CTR
Record Dates: First submitted 2014-05-12; First posted 2014-05-13 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-08

CONDITIONS: Type 1 Diabetes
Keywords: Artificial Pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Closed-Loop Control System (Experimental): Use of an investigational control-to-range automated insulin management (artificial pancreas) system using continuous glucose monitoring (CGM) and subcutaneous insulin pump infusion in individuals with type 1 diabetes in the home environment.
  Interventions: Device: Closed-Loop Control System
- Sensor-Augmented Pump (SAP) (Active Comparator): Use of a study-assigned commercial continuous glucose monitoring (CGM) system and commercial insulin pump
  Interventions: Device: Sensor-Augmented Pump (SAP)

INTERVENTIONS:
Device: Closed-Loop Control System — This investigational device system included the following components:
  * DiAs - a smart-phone medical platform;
  * Dexcom G4 Platinum CGM system connected to DiAs via CGM receiver and USB-Bluetooth relay hardware;
  * Roche Accu-Chek insulin pump connected to DiAs via wireless Bluetooth;
  * Remote Monitoring Server connected to DiAs via 3G or local Wi-Fi network
  * Modular Closed-Loop Control Algorithm Running on DiAs, which is of Control-to-Range (CTR) class
  Other Names: Diabetes Assistant (DiAs)
  Arms: Closed-Loop Control System
Device: Sensor-Augmented Pump (SAP) — This commercial device system included the following components:
  * Dexcom G4 Platinum CGM system;
  * Roche Accu-Chek insulin pump
  Arms: Sensor-Augmented Pump (SAP)

SUMMARY:
The purpose of this study is to see if an automated insulin management system ("study system") can safely be used at home to manage blood sugar. The study system includes (1) a CGM that measures glucose levels, (2) a computer program on a smartphone that determines how much insulin is needed and allows the study participant user to control the whole system, and (3) an insulin pump that delivers the insulin. The CGM will be from Dexcom. The pump will be from Roche. The CGM and pump are similar to the devices that are currently available for people to purchase and use. However, the smartphone device, the CGM sensor type used with it, and the overall study system can only be used for research at this time.

The study will be completed by about 24 individuals at 6 centers in the United States and Europe. This study has several phases and will take about 11-14 weeks to complete depending on whether the study participant is a CGM user or not.

At selected sites (based on subject eligibility and availability), approximately 10-20 subjects who exhibit safe and competent use of the system at home will be given the option to continue home use of the system in Day-and-Night Closed-Loop mode for up to 5 months.

DETAILED DESCRIPTION:
The study phases are as follows:

* Screening visit to see if you are eligible for the study and to determine how long you will need to use the study CGM (visit 1)
* Up to 3 weeks using the study CGM (depends on your current CGM use), followed by an office visit (visit 2)
* 2 weeks using the study insulin pump and study CGM together
* Full day visit in clinic or hotel for training using the system (visit 3)
* 1 week using the system without automated insulin delivery or suspension
* 2-day hotel or clinic visit for closed-loop training (visit 4),
* 16-19 days using the system in the evening and overnight only followed by an office visit (visit 5)
* 16-19 days using the system for the full 24 hours
* Final study clinic visit (visit 6)
* Option 5 month extension phase of day-and-night closed-loop home use

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year and using insulin for at least 1 year and an insulin pump for at least 6 months.
2. Age >=18 to <70 years.
3. HbA1c <10.0%; if HbA1c <6.0% then total daily insulin must be >=0.5 U/kg
4. For females, not currently known to be pregnant. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative urine pregnancy test will be required for all premenopausal women who are not surgically sterile. Subjects who become pregnant will be discontinued from the study.
5. Demonstration of proper mental status and cognition for the study.
6. Currently using insulin-to-carbohydrate ratio to calculate meal bolus sizes
7. Hypoglycemia awareness as demonstrated by a Clarke Hypoglycemia Awareness score of 2 or lower
8. Access to internet and cell phone service at home, and a computer for downloading device data.
9. Living with significant other or family member committed to participating in all training activities, knowledgeable at all times of the participant's location, and being present and available to provide assistance when system is being used at night.
10. Commitment to maintaining uninterrupted availability via cell phone and avoiding any overnight travel for the duration of each two-week period using the closed-loop system.
11. An understanding of and willingness to follow the protocol and sign the informed consent.

Exclusion Criteria:

1. Admission for diabetic ketoacidosis in the 12 months prior to enrollment.
2. Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment.
3. History of a seizure disorder (except hypoglycemic seizure), unless written clearance is received from a neurologist.
4. Coronary artery disease or heart failure, unless written clearance is received from a cardiologist.
5. History of cardiac arrhythmia (except for benign premature atrial contractions and benign premature ventricular contractions which are permitted)
6. Cystic fibrosis.
7. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:

   * Inpatient psychiatric treatment in the past 6 months for either the subject or the subject's primary care giver (i.e., parent or guardian)
   * Presence of a known adrenal disorder
   * Abnormal liver function test results (Transaminase >2 times the upper limit of normal); testing required for subjects taking medications known to affect liver function or with diseases known to affect liver function
   * Abnormal renal function test results (calculated GFR <60); testing required for subjects with diabetes duration of greater than 5 years post onset of puberty
   * Active gastroparesis
   * If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
   * Uncontrolled thyroid disease (TSH undetectable or >10); testing required within three months prior to admission for subjects with a goiter, positive antibodies, or who are on thyroid hormone replacement, and within one year otherwise
   * Abuse of alcohol or recreational drugs
   * Infectious process not anticipated to resolve prior to study procedures (e.g. meningitis, pneumonia, osteomyelitis)

7. A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the protocol 8. Current use of the following drugs and supplements:

* Acetaminophen
* Any medication being taken to lower blood glucose, such as Pramlintide, Metformin, GLP-1 Analogs such as Liraglutide, and nutraceuticals intended to lower blood glucose
* Beta blockers
* Oral or injectable glucocorticoids
* Any other medication that the investigator believes is a contraindication to the subject's participation

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Beck, MD, PhD, Principal Investigator — Jaeb Center for Health Research; Boris Kovatchev, PhD, Study Chair — University of Virginia
Locations (6):
- United States (3):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Stanford University, Stanford, California
  - University of Virginia, Charlottesville, Virginia
- Montpellier University Hospital, Montpellier, France
- National Center for Childhood Diabetes- Schneider Children's Medical Center, Petah Tikva, Israel
- University of Padova, Padua, Italy

REFERENCES:
- [Result] Anderson SM, Raghinaru D, Pinsker JE, Boscari F, Renard E, Buckingham BA, Nimri R, Doyle FJ 3rd, Brown SA, Keith-Hynes P, Breton MD, Chernavvsky D, Bevier WC, Bradley PK, Bruttomesso D, Del Favero S, Calore R, Cobelli C, Avogaro A, Farret A, Place J, Ly TT, Shanmugham S, Phillip M, Dassau E, Dasanayake IS, Kollman C, Lum JW, Beck RW, Kovatchev B; Control to Range Study Group. Multinational Home Use of Closed-Loop Control Is Safe and Effective. Diabetes Care. 2016 Jul;39(7):1143-50. doi: 10.2337/dc15-2468. Epub 2016 Apr 13. PMID 27208316
- See also: Multinational Home Use of Closed-Loop Control Is Safe and Effective — https://www.ncbi.nlm.nih.gov/pubmed/27208316

RESULTS

PARTICIPANT FLOW:
Groups:
- Closed-Loop Control System: A control-to-range automated insulin management system using continuous glucose monitoring (CGM) and subcutaneous insulin pump infusion in individuals with type 1 diabetes in the home environment.
  Closed-Loop Control System: The devices that will be used in the Closed-Loop Control System include the following components:
  * DiAs - a smart-phone medical platform;
  * Dexcom Dexcom G4 Platinum connected to DiAs via CGM receiver and USB-Bluetooth relay hardware;
  * Roche Accu-Chek insulin pump connected to DiAs via wireless Bluetooth;
  * Remote Monitoring Server connected to DiAs via 3G or local Wi-Fi network, and
  * Modular Closed-Loop Control Algorithm Running on DiAs, which is of Control-to-Range (CTR) class
Period: 2-Week Baseline Sensor-Augmented Pump
Arm/Group | Closed-Loop Control System
Started | 30
Completed | 30
Not Completed | 0
Period: 2-Week Overnight-Only Closed-Loop
Arm/Group | Closed-Loop Control System
Started | 30
Completed | 30
Not Completed | 0
Period: 2-Week 24/7 Closed-Loop
Arm/Group | Closed-Loop Control System
Started | 30
Completed | 30
Not Completed | 0
Period: 5-Month 24/7 Closed-Loop
Arm/Group | Closed-Loop Control System
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Closed-Loop Control System
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 44 [18 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 15
  Italy | 5
  Israel | 5
  France | 5
Diabetes duration [Median (Inter-Quartile Range); unit: years] | 19 [13 to 28]
Body-mass index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 25 [23 to 27]
Hemoglobin A1c (HbA1c) [Median (Inter-Quartile Range); unit: percent] | 7.3 [7.1 to 7.7]
Daily total insulin dose [Median (Inter-Quartile Range); unit: U/kg/day] | 0.57 [0.42 to 0.72]
Daily basal insulin [Median (Inter-Quartile Range); unit: U/kg/day] | 0.27 [0.20 to 0.37]

OUTCOME MEASURES:

1. Primary Outcome: Time Spent <70 mg/dL - Main Phase, Night Only
Description: Percentage of CGM Measured Glucose Values <70 mg/dl during study Main Phase, night only (23:00 to 07:00)
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Groups:
- 2-Week Baseline Sensor-Augmented Pump: Home use of a study-assigned commercial continuous glucose monitoring (CGM) system and commercial insulin pump for a 2-Week period
- 2-Week Overnight-Only Closed-Loop: Overnight-only home use of a control-to-range automated insulin management system using continuous glucose monitoring (CGM) and subcutaneous insulin pump infusion in individuals with type 1 diabetes for a 2-Week period
- 2-Week 24/7 Closed-Loop: 24/7 (night and day) home use of a control-to-range automated insulin management system using continuous glucose monitoring (CGM) and subcutaneous insulin pump infusion in individuals with type 1 diabetes for a 2-Week period
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 3.0 [1.1 to 6.3] | 1.1 [0.2 to 1.6] | 0.4 [0.2 to 1.7]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority — No adjustments were made for multiple comparisons; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.31, t-test, 2 sided — No adjustments were made for multiple comparisons

2. Secondary Outcome: Time Spent <70 mg/dL - Main Phase, Day and Night
Description: Percentage of CGM Measured Glucose Values <70 mg/dl during study Main Phase
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 4.1 [2.0 to 7.8] | 2.6 [1.6 to 3.6] | 1.7 [1.1 to 2.7]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.002, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons

3. Secondary Outcome: Time Spent <70 mg/dL - Main Phase, Day Only
Description: Percentage of CGM Measured Glucose Values <70 mg/dl during study Main Phase, day only (07:00 - 23:00)
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 4.6 [2.0 to 7.0] | 3.2 [2.1 to 4.6] | 2.3 [1.3 to 3.0]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.10, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons

4. Secondary Outcome: Time in Range 70-180 mg/dL - Main Phase, Day and Night
Description: Percentage of CGM Measured Glucose Values in range 70-180 mg/dl during study Main Phase
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 65 [59 to 69] | 73 [65 to 78] | 73 [68 to 76]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.91, t-test, 2 sided — No adjustments were made for multiple comparisons

5. Secondary Outcome: Time in Range 70-180 mg/dL - Main Phase, Night Only
Description: Percentage of CGM Measured Glucose Values in range 70-180 mg/dl during study Main Phase, night only (23:00 - 07:00)
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 61 [53 to 73] | 75 [69 to 80] | 72 [65 to 80]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.20, t-test, 2 sided — No adjustments were made for multiple comparisons

6. Secondary Outcome: Time in Range 70-180 mg/dL - Main Phase, Day Only
Description: Percentage of CGM Measured Glucose Values in range 70-180 mg/dl during study Main Phase, day only (07:00 - 23:00)
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 65 [61 to 71] | 70 [65 to 77] | 72 [69 to 78]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.49, t-test, 2 sided — No adjustments were made for multiple comparisons

7. Secondary Outcome: Mean Sensor Glucose - Main Phase, Day and Night
Description: Mean CGM sensor glucose during study Main Phase
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
mg/dL | 157 (18) | 149 (12) | 153 (12)
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.009, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.14, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.06, t-test, 2 sided — No adjustments were made for multiple comparisons

8. Secondary Outcome: Mean Sensor Glucose - Main Phase, Night Only
Description: Mean CGM sensor glucose during study Main Phase, night only (23:00 - 07:00)
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
mg/dL | 163 (23) | 150 (12) | 154 (13)
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.002, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.03, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.18, t-test, 2 sided — No adjustments were made for multiple comparisons

9. Secondary Outcome: Mean Sensor Glucose - Main Phase, Day Only
Description: Mean CGM sensor glucose during study Main Phase, day only (07:00 - 23:00)
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
mg/dL | 154 (19) | 148 (15) | 152 (14)
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.07, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.54, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.07, t-test, 2 sided — No adjustments were made for multiple comparisons

10. Secondary Outcome: Glucose Coefficient of Variation - Main Phase, Day and Night
Description: CGM Glucose Coefficient of Variation (CV) during study Main Phase
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage | 38 [34 to 41] | 35 [33 to 37] | 34 [31 to 37]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.005, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.02, t-test, 2 sided — No adjustments were made for multiple comparisons

11. Secondary Outcome: Glucose Coefficient of Variation - Main Phase, Night Only
Description: CGM Glucose Coefficient of Variation (CV) during study Main Phase, night only (23:00 - 07:00)
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage | 36 [32 to 40] | 30 [29 to 34] | 32 [27 to 36]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.52, t-test, 2 sided — No adjustments were made for multiple comparisons

12. Secondary Outcome: Glucose Coefficient of Variation - Main Phase, Day Only
Description: CGM Glucose Coefficient of Variation (CV) during study Main Phase, day only (07:00 - 23:00)
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage | 38 [34 to 42] | 37 [34 to 39] | 35 [31 to 37]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.13, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons

13. Secondary Outcome: Glucose Standard Deviation - Main Phase, Day and Night
Description: CGM Glucose Standard Deviation (SD) during study Main Phase
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
mg/dL | 61 [53 to 69] | 52 [48 to 58] | 51 [47 to 55]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.41, t-test, 2 sided — No adjustments were made for multiple comparisons

14. Secondary Outcome: Glucose Standard Deviation - Main Phase, Night Only
Description: CGM Glucose Standard Deviation (SD) during study Main Phase, night only (23:00 - 07:00)
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
mg/dL | 61 [50 to 69] | 47 [42 to 51] | 48 [40 to 58]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.12, t-test, 2 sided — No adjustments were made for multiple comparisons

15. Secondary Outcome: Glucose Standard Deviation - Main Phase, Day Only
Description: CGM Glucose Standard Deviation (SD) during study Main Phase, day only (07:00 - 23:00)
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
mg/dL | 58 [53 to 65] | 55 [49 to 60] | 53 [47 to 54]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.02, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.06, t-test, 2 sided — No adjustments were made for multiple comparisons

16. Secondary Outcome: Time Spent >180 mg/dL - Main Phase, Day and Night
Description: Percentage of CGM Measured Glucose Values >180 mg/dl during study Main Phase
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 32 [25 to 36] | 24 [20 to 31] | 25 [22 to 28]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.26, t-test, 2 sided — No adjustments were made for multiple comparisons

17. Secondary Outcome: Time Spent >180 mg/dL - Main Phase, Night Only
Description: Percentage of CGM Measured Glucose Values >180 mg/dl during study Main Phase, night only (23:00 to 07:00)
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 37 [24 to 45] | 24 [19 to 28] | 27 [19 to 34]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.11, t-test, 2 sided — No adjustments were made for multiple comparisons

18. Secondary Outcome: Time Spent >180 mg/dL - Main Phase, Day Only
Description: Percentage of CGM Measured Glucose Values >180 mg/dl during study Main Phase, day only (07:00 - 23:00)
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 31 [23 to 35] | 23 [19 to 32] | 25 [21 to 29]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.02, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.02, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.61, t-test, 2 sided — No adjustments were made for multiple comparisons

19. Secondary Outcome: Time Spent <50 mg/dL - Main Phase, Day and Night
Description: Percentage of CGM Measured Glucose Values <50 mg/dl during study Main Phase
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 0.8 [0.1 to 1.3] | 0.2 [0.1 to 0.5] | 0.2 [0.0 to 0.4]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.29, t-test, 2 sided — No adjustments were made for multiple comparisons

20. Secondary Outcome: Time Spent <50 mg/dL - Main Phase, Night Only
Description: Percentage of CGM Measured Glucose Values <50 mg/dl during study Main Phase, night only (23:00 to 07:00)
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 0.3 [0.0 to 1.0] | 0.0 [0.0 to 0.1] | 0.0 [0.0 to 0.1]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.005, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p > 0.99, t-test, 2 sided — No adjustments were made for multiple comparisons

21. Secondary Outcome: Time Spent <50 mg/dL - Main Phase, Day Only
Description: Percentage of CGM Measured Glucose Values <50 mg/dl during study Main Phase, day only (07:00 - 23:00)
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 0.9 [0.1 to 1.2] | 0.2 [0.1 to 0.7] | 0.2 [0.0 to 0.4]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.006, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.09, t-test, 2 sided — No adjustments were made for multiple comparisons

22. Secondary Outcome: Time Spent <60 mg/dL - Main Phase, Day and Night
Description: Percentage of CGM Measured Glucose Values <60 mg/dl during study Main Phase
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 2.2 [0.7 to 3.5] | 1.1 [0.5 to 1.5] | 0.7 [0.3 to 1.0]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.002, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons

23. Secondary Outcome: Time Spent <60 mg/dL - Main Phase, Night Only
Description: Percentage of CGM Measured Glucose Values <60 mg/dl during study Main Phase, night only (23:00 - 07:00)
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 1.4 [0.4 to 2.9] | 0.2 [0.0 to 0.6] | 0.1 [0.0 to 0.6]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.26, t-test, 2 sided — No adjustments were made for multiple comparisons

24. Secondary Outcome: Time Spent <60 mg/dL - Main Phase, Day Only
Description: Percentage of CGM Measured Glucose Values <60 mg/dl during study Main Phase, day only (07:00 - 23:00)
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 2.4 [0.8 to 3.5] | 1.4 [0.7 to 1.9] | 0.7 [0.4 to 1.1]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.04, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons

25. Secondary Outcome: LBGI - Main Phase, Day and Night
Description: Low Blood Glucose Index (LBGI) - Main Phase, Day and Night. The LGBI metric is used to quantify the risk of hypoglycemia. A higher LBGI implies more mild hypoglycemic events or less severe hypoglycemic events.
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: index scores
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
index scores | 1.1 [0.6 to 1.9] | 0.8 [0.6 to 0.9] | 0.6 [0.4 to 0.8]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.006, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons

26. Secondary Outcome: LBGI - Main Phase, Night Only
Description: Low Blood Glucose Index (LBGI) - Main Phase, night only (23:00 - 07:00). The LGBI metric is used to quantify the risk of hypoglycemia. A higher LBGI implies more mild hypoglycemic events or less severe hypoglycemic events.
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: index scores
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
index scores | 0.7 [0.4 to 1.6] | 0.4 [0.3 to 0.5] | 0.3 [0.2 to 0.6]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p < 0.001, t-test, 1 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.53, t-test, 2 sided — No adjustments were made for multiple comparisons

27. Secondary Outcome: LBGI - Main Phase, Day Only
Description: Low Blood Glucose Index (LBGI) - Main Phase, day only (07:00 - 23:00). The LGBI metric is used to quantify the risk of hypoglycemia. A higher LBGI implies more mild hypoglycemic events or less severe hypoglycemic events.
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: index scores
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
index scores | 1.2 [0.8 to 1.7] | 0.9 [0.7 to 1.2] | 0.7 [0.4 to 0.9]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.05, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons

28. Secondary Outcome: AOC 70 mg/dL - Main Phase, Day and Night
Description: Area Over the Curve (AOC) 70 mg/dL - Main Phase, Day and Night. The hypoglycemia AOC is scaled to the number of CGM readings so the time factor cancels out. Technically, the units would be mg/dl, but this might seem unintuitive since it is incremental relative to a threshold. For example, a hypoglycemia AOC of 1 mg/dl can denote a glucose of 60 mg/dl for 10% of the time (10 mg/dl below threshold * 10% = 1 mg/dl) or 65 mg/dl for 20% of the time (5 mg/dl below threshold * 20% = 1 mg/dl). Note that it is based on relative (%) rather than absolute time so there is no time element in the resulting units.
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
mg/dL | 0.5 [0.2 to 0.9] | 0.3 [0.1 to 0.4] | 0.2 [0.1 to 0.3]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons

29. Secondary Outcome: AOC 70 mg/dL - Main Phase, Night Only
Description: Area Over the Curve (AOC) 70 mg/dL - Main Phase, night only (23:00 - 07:00). The hypoglycemia AOC is scaled to the number of CGM readings so the time factor cancels out. Technically, the units would be mg/dl, but this might seem unintuitive since it is incremental relative to a threshold. For example, a hypoglycemia AOC of 1 mg/dl can denote a glucose of 60 mg/dl for 10% of the time (10 mg/dl below threshold * 10% = 1 mg/dl) or 65 mg/dl for 20% of the time (5 mg/dl below threshold * 20% = 1 mg/dl). Note that it is based on relative (%) rather than absolute time so there is no time element in the resulting units.
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
mg/dL | 0.3 [0.1 to 0.6] | 0.1 [0.0 to 0.2] | 0.0 [0.0 to 0.2]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.22, t-test, 2 sided — No adjustments were made for multiple comparisons

30. Secondary Outcome: AOC 70 mg/dL - Main Phase, Day Only
Description: Area Over the Curve (AOC) 70 mg/dL - Main Phase, day only (07:00 - 23:00). The hypoglycemia AOC is scaled to the number of CGM readings so the time factor cancels out. Technically, the units would be mg/dl, but this might seem unintuitive since it is incremental relative to a threshold. For example, a hypoglycemia AOC of 1 mg/dl can denote a glucose of 60 mg/dl for 10% of the time (10 mg/dl below threshold * 10% = 1 mg/dl) or 65 mg/dl for 20% of the time (5 mg/dl below threshold * 20% = 1 mg/dl). Note that it is based on relative (%) rather than absolute time so there is no time element in the resulting units.
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
mg/dL | 0.6 [0.2 to 0.9] | 0.3 [0.2 to 0.5] | 0.2 [0.1 to 0.3]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.03, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons

31. Secondary Outcome: HBGI - Main Phase, Day and Night
Description: High Blood Glucose Index (HBGI) - Main Phase, Day and Night. The HBGI metric is used to quantify the risk of hyperglycemia. A higher HBGI implies more mild hyperglycemic events or less severe hyperglycemic events.
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: index scores
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
index scores | 6.8 [5.9 to 7.8] | 5.0 [4.3 to 6.2] | 5.5 [4.6 to 6.7]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.26, t-test, 2 sided — No adjustments were made for multiple comparisons

32. Secondary Outcome: HBGI - Main Phase, Night Only
Description: High Blood Glucose Index (HBGI) - Main Phase, night only (23:00 - 07:00). The HBGI metric is used to quantify the risk of hyperglycemia. A higher HBGI implies more mild hyperglycemic events or less severe hyperglycemic events.
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: index scores
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
index scores | 7.5 [5.4 to 9.7] | 5.1 [4.1 to 5.7] | 5.4 [4.3 to 6.7]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.05, t-test, 2 sided — No adjustments were made for multiple comparisons

33. Secondary Outcome: HBGI - Main Phase, Day Only
Description: High Blood Glucose Index (HBGI) - Main Phase, day only (07:00 - 23:00). The HBGI metric is used to quantify the risk of hyperglycemia. A higher HBGI implies more mild hyperglycemic events or less severe hyperglycemic events.
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: index scores
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
index scores | 6.4 [5.2 to 8.0] | 5.1 [4.4 to 7.1] | 5.5 [4.7 to 6.3]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.03, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.02, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.52, t-test, 2 sided — No adjustments were made for multiple comparisons

34. Secondary Outcome: ADRR - Main Phase, Day and Night
Description: Average Daily Risk Range (ADRR) - Main Phase, Day and Night. ADRR is a metric that categorizes risk for hyper and hypoglycemic events. Low risk is scored 0-19, moderate risk is scored 20-40, and high risk is 40 and above.
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: range scores
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
range scores | 27 [25 to 34] | 24 [21 to 28] | 24 [19 to 27]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.003, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.71, t-test, 2 sided — No adjustments were made for multiple comparisons

35. Secondary Outcome: AUC 180 mg/dL - Main Phase, Day and Night
Description: Area Under the Curve (AUC) 180 mg/dL - Main Phase, Day and Night. The hyperglycemic AUC is scaled to the number of CGM readings so the time factor cancels out. Technically, the units would be mg/dl, but this might seem unintuitive since it is incremental relative to a threshold. For example, the hyperglycemic AUC is 28 (mg/dl)*days for Patient A and 56 (mg/dl)*days for Patient B when using 180 as the threshold. But this is artificial because Patient B wore the sensor twice as long. So we similarly scale it relative to the number of readings to reflect a mean rather than a sum. So we say hyperglycemic AUC = 4 mg/dl for both patients. Note that time disappears from the units in the scaled version. It represents the mean value of max(glucose-180, 0).
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
mg/dL | 15.0 [11.7 to 18.4] | 9.2 [7.7 to 13.4] | 11.3 [7.6 to 14.2]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.39, t-test, 2 sided — No adjustments were made for multiple comparisons

36. Secondary Outcome: AUC 180 mg/dL - Main Phase, Night Only
Description: Area Under the Curve (AUC) 180 mg/dL - Main Phase, night only (23:00 - 07:00). The hyperglycemic AUC is scaled to the number of CGM readings so the time factor cancels out. Technically, the units would be mg/dl, but this might seem unintuitive since it is incremental relative to a threshold. For example, the hyperglycemic AUC is 28 (mg/dl)*days for Patient A and 56 (mg/dl)*days for Patient B when using 180 as the threshold. But this is artificial because Patient B wore the sensor twice as long. So we similarly scale it relative to the number of readings to reflect a mean rather than a sum. So we say hyperglycemic AUC = 4 mg/dl for both patients. Note that time disappears from the units in the scaled version. It represents the mean value of max(glucose-180, 0).
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
mg/dL | 17.7 [7.9 to 26.4] | 8.4 [5.7 to 11.0] | 9.1 [6.4 to 14.2]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.06, t-test, 2 sided — No adjustments were made for multiple comparisons

37. Secondary Outcome: AUC 180 mg/dL - Main Phase, Day Only
Description: Area Under the Curve (AUC) 180 mg/dL - Main Phase, day only (07:00 - 23:00). The hyperglycemic AUC is scaled to the number of CGM readings so the time factor cancels out. Technically, the units would be mg/dl, but this might seem unintuitive since it is incremental relative to a threshold. For example, the hyperglycemic AUC is 28 (mg/dl)*days for Patient A and 56 (mg/dl)*days for Patient B when using 180 as the threshold. But this is artificial because Patient B wore the sensor twice as long. So we similarly scale it relative to the number of readings to reflect a mean rather than a sum. So we say hyperglycemic AUC = 4 mg/dl for both patients. Note that time disappears from the units in the scaled version. It represents the mean value of max(glucose-180, 0).
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
mg/dL | 13.6 [9.6 to 17.9] | 10.0 [7.7 to 15.3] | 9.8 [7.5 to 14.0]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.02, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.003, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.86, t-test, 2 sided — No adjustments were made for multiple comparisons

38. Secondary Outcome: Time Spent >250 mg/dL - Main Phase, Day and Night
Description: Percentage of CGM Measured Glucose Values >250 mg/dl during study Main Phase
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 7 [4 to 11] | 4 [3 to 7] | 5 [3 to 7]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.74, t-test, 2 sided — No adjustments were made for multiple comparisons

39. Secondary Outcome: Time Spent >250 mg/dL - Main Phase, Night Only
Description: Percentage of CGM Measured Glucose Values >250 mg/dl during study Main Phase, night only (23:00 to 07:00)
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 8 [3 to 14] | 3 [2 to 6] | 4 [2 to 6]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.09, t-test, 2 sided — No adjustments were made for multiple comparisons

40. Secondary Outcome: Time Spent >250 mg/dL - Main Phase, Day Only
Description: Percentage of CGM Measured Glucose Values >250 mg/dl during study Main Phase, day only (07:00 - 23:00)
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 6 [3 to 10] | 5 [3 to 6] | 5 [3 to 7]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.07, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.006, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.68, t-test, 2 sided — No adjustments were made for multiple comparisons

41. Secondary Outcome: Time Spent >300 mg/dL - Main Phase, Day and Night
Description: Percentage of CGM Measured Glucose Values >300 mg/dl during study Main Phase
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 2 [1 to 3] | 1 [0 to 2] | 1 [0 to 2]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.006, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.005, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.62, t-test, 2 sided — No adjustments were made for multiple comparisons

42. Secondary Outcome: Time Spent >300 mg/dL - Main Phase, Night Only
Description: Percentage of CGM Measured Glucose Values >300 mg/dl during study Main Phase, night only (23:00 to 07:00)
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 2 [0 to 6] | 0 [0 to 1] | 0 [0 to 2]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.006, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.23, t-test, 2 sided — No adjustments were made for multiple comparisons

43. Secondary Outcome: Time Spent >300 mg/dL - Main Phase, Day Only
Description: Percentage of CGM Measured Glucose Values >300 mg/dl during study Main Phase, day only (07:00 - 23:00)
Time Frame: 2 weeks
Population: One participant was excluded due to missing baseline CGM data
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 2-Week Overnight-Only Closed-Loop | 2-Week 24/7 Closed-Loop
Number analyzed (Participants) | 29 | 29 | 29
percentage of CGM values | 2 [0 to 3] | 1 [1 to 2] | 1 [0 to 2]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week Overnight-Only Closed-Loop; Test type: Superiority; p = 0.67, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.09, t-test, 2 sided — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: 2-Week Overnight-Only Closed-Loop vs 2-Week 24/7 Closed-Loop; Test type: Superiority; p = 0.22, t-test, 2 sided — No adjustments were made for multiple comparisons

44. Other Pre Specified Outcome: Mean Sensor Glucose - Extension Phase
Description: Mean CGM sensor glucose during Extension Phase
Time Frame: 3 months
Population: One subject had missing CGM data at baseline and was not included in this analysis
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- 5-Month 24/7 Closed-Loop: 24/7 (night and day) home use of a control-to-range automated insulin management system using continuous glucose monitoring (CGM) and subcutaneous insulin pump infusion in individuals with type 1 diabetes for a 5-Month period
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 5-Month 24/7 Closed-Loop
Number analyzed (Participants) | 13 | 13
mmol/L | 8.6 (1.1) | 8.3 (0.6)
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 5-Month 24/7 Closed-Loop; Test type: Superiority; p = 0.25, t-test, 2 sided — No adjustments were made for multiple comparisons

45. Other Pre Specified Outcome: Change in HbA1c - Extension Phase
Description: Comparison of HbA1c collected at baseline and at the end of the 5-month extension phase
Time Frame: 5 months
Population: One participant was excluded due to missing baseline CGM data
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 5-Month 24/7 Closed-Loop
Number analyzed (Participants) | 13 | 13
percentage | 7.2 (0.6) | 7.0 (0.6)
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 5-Month 24/7 Closed-Loop; Test type: Superiority; p = 0.23, t-test, 2 sided — No adjustments were made for multiple comparisons

46. Other Pre Specified Outcome: Time Spent <3.9 mmol/L (70 mg/dL) - Extension Phase
Description: Percentage of CGM Measured Glucose Values <3.9 mmol/L (70 mg/dL) during study Extension Phase
Time Frame: 3 months
Population: One subject had missing CGM data at baseline and was not included in this analysis
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 5-Month 24/7 Closed-Loop
Number analyzed (Participants) | 13 | 13
mmol/L | 4.1 [2.9 to 7.5] | 1.3 [0.6 to 1.7]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 5-Month 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons

47. Other Pre Specified Outcome: Time Spent <3.3 mmol/L (60 mg/dL) - Extension Phase
Description: Percentage of CGM Measured Glucose Values <3.3 mmol/L (60 mg/dL) during study Extension Phase
Time Frame: 3 months
Population: One subject had missing CGM data at baseline and was not included in this analysis
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 5-Month 24/7 Closed-Loop
Number analyzed (Participants) | 13 | 13
mmol/L | 2.2 [1.5 to 3.4] | 0.3 [0.2 to 0.6]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 5-Month 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons

48. Other Pre Specified Outcome: Time Spent <2.8 mmol/L (50 mg/dL) - Extension Phase
Description: Percentage of CGM Measured Glucose Values <2.8 mmol/L (50 mg/dL) during study Extension Phase
Time Frame: 3 months
Population: One subject had missing CGM data at baseline and was not included in this analysis
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 5-Month 24/7 Closed-Loop
Number analyzed (Participants) | 13 | 13
mmol/L | 1.0 [0.8 to 1.3] | 0.1 [0.0 to 0.2]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 5-Month 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons

49. Other Pre Specified Outcome: Time in Range 3.9-10.0 mmol/L (70-180 mg/dL) - Extension Phase
Description: Percentage of CGM Measured Glucose Values in range 3.9-10.0 mmol/L (70-180 mg/dL)
Time Frame: 3 months
Population: One subject had missing CGM data at baseline and was not included in this analysis
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values in range
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 5-Month 24/7 Closed-Loop
Number analyzed (Participants) | 13 | 13
percentage of CGM values in range | 66 [59 to 69] | 77 [73 to 81]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 5-Month 24/7 Closed-Loop; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments were made for multiple comparisons

50. Other Pre Specified Outcome: Time Spent >10.0 mmol/L (180 mg/dL) - Extension Phase
Description: Percentage of CGM Measured Glucose Values >10.0 mmol/L (180 mg/dL) during study Extension Phase
Time Frame: 3 months
Population: One subject had missing CGM data at baseline and was not included in this analysis
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values >10.0 mmol/L
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 5-Month 24/7 Closed-Loop
Number analyzed (Participants) | 13 | 13
percentage of CGM values >10.0 mmol/L | 31 [23 to 38] | 22 [19 to 27]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 5-Month 24/7 Closed-Loop; Test type: Superiority; p = 0.01, t-test, 2 sided — No adjustments were made for multiple comparisons

51. Other Pre Specified Outcome: Time Spent >13.9 mmol/L (250 mg/dL) - Extension Phase
Description: Percentage of CGM Measured Glucose Values >13.9 mmol/L (250 mg/dL) during study Extension Phase
Time Frame: 3 months
Population: One subject had missing CGM data at baseline and was not included in this analysis
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values in range
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 5-Month 24/7 Closed-Loop
Number analyzed (Participants) | 13 | 13
percentage of CGM values in range | 6 [3 to 11] | 3 [2 to 6]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 5-Month 24/7 Closed-Loop; Test type: Superiority; p = 0.006, t-test, 2 sided — No adjustments were made for multiple comparisons

52. Other Pre Specified Outcome: Time Spent >16.7 mmol/L (300 mg/dL) - Extension Phase
Description: Percentage of CGM Measured Glucose Values >16.7 mmol/L (300 mg/dL) during study Extension Phase
Time Frame: 3 months
Population: One subject had missing CGM data at baseline and was not included in this analysis
Measure: Median (Inter-Quartile Range); unit: percentage of CGM values in range
Arm/Group | 2-Week Baseline Sensor-Augmented Pump | 5-Month 24/7 Closed-Loop
Number analyzed (Participants) | 13 | 13
percentage of CGM values in range | 2 [0 to 3] | 0 [0 to 1]
Statistical Analysis 1: Comparison: 2-Week Baseline Sensor-Augmented Pump vs 5-Month 24/7 Closed-Loop; Test type: Superiority; p = 0.14, t-test, 2 sided — No adjustments were made for multiple comparisons

53. Other Pre Specified Outcome: Episodes of Severe Hypoglycemia Events - Extension Phase
Description: Episodes of severe hypoglycemia events during the 5-month extension phase defined as an event requiring assistance of another person due to altered consciousness to actively administer carbohydrate, glucagon, or other resuscitative actions. This means that the subject was impaired cognitively to the point that he/she was unable to treat him or herself, was unable to verbalize his or her needs, was incoherent, disoriented, and/or combative, or experienced seizure or coma. These episodes may be associated with sufficient neuroglycopenia to induce seizure or coma. If plasma glucose measurements are not available during such an event, neurological recovery attributable to the restoration of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration.
Time Frame: 5 months
Measure: Number; unit: events
Arm/Group | 5-Month 24/7 Closed-Loop
Number analyzed (Participants) | 14
events | 0

54. Other Pre Specified Outcome: Episodes of Diabetic Ketoacidosis (DKA) Events - Extension Phase
Description: Episodes of DKA events that occurred during the 5-month extension phase
Time Frame: 5 months
Measure: Number; unit: events
Arm/Group | 5-Month 24/7 Closed-Loop
Number analyzed (Participants) | 14
events | 0

55. Other Pre Specified Outcome: Reported Serious Adverse Events - Extension Phase
Description: Reported serious adverse events during the 5-month extension phase
Time Frame: 5 months
Measure: Number; unit: events
Arm/Group | 5-Month 24/7 Closed-Loop
Number analyzed (Participants) | 14
events | 0

ADVERSE EVENTS:
Time Frame: 12-weeks during the main portion of the study and 5 months in the optional extension phase of the study.
Arm/Group | Closed-Loop Control System
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 9/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Closed-Loop Control System (N=30)
Urinary tract infection (Renal and urinary disorders) | 1 (2) — Was assessed by site principal investigator and study medical monitor as unrelated to study device and/or procedure.
Endometriosis (Reproductive system and breast disorders) | 1 (1) — Was assessed by site principal investigator and study medical monitor as unrelated to study device and/or procedure.
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Was assessed by site principal investigator and study medical monitor as unrelated to study device and/or procedure.
Cold (General disorders) | 2 (2) — Was assessed by site principal investigator and study medical monitor as unrelated to study device and/or procedure.
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Was assessed by site principal investigator and study medical monitor as unrelated to study device and/or procedure.
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Was assessed by site principal investigator and study medical monitor as unrelated to study device and/or procedure.
Ketosis (Endocrine disorders) | 1 (2)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Was assessed by site principal investigator and study medical monitor as unrelated to study device and/or procedure.
Tooth Infection (Infections and infestations) | 1 (1) — Was assessed by site principal investigator and study medical monitor as unrelated to study device and/or procedure.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Was assessed by site principal investigator and study medical monitor as unrelated to study device and/or procedure.
Skin injury (Injury, poisoning and procedural complications) | 1 (1) — Was assessed by site principal investigator and study medical monitor as unrelated to study device and/or procedure.
Hyperglycemia (Endocrine disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) — Was assessed by site principal investigator and study medical monitor as unrelated to study device and/or procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No